CLINICAL TRIAL: NCT06215963
Title: App for Independence-O (A4i-O) - Expanding a Validated Platform for Complex Behavioral Health to Address Opioid Use Disorder
Brief Title: A4i-O: A Platform for Complex Behavioral Health to Address OUD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Sean Kidd, Senior Scientist, Centre for Addiction and Mental Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 042/2022
Record Dates: First submitted 2023-12-12; First posted 2024-01-22 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-01

CONDITIONS: Opioid-Related Disorders; Relationship, Professional Patient; Mental Health Wellness 1; Mobile Phone Use; Comorbidities and Coexisting Conditions
Keywords: Opioid Use Disorder; Digital Health Intervention; Substance Use; Mental Health and Wellness
MeSH Terms: conditions — Opioid-Related Disorders; Cell Phone Use; Substance-Related Disorders; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- App for Independence-O (A4i-O) (Experimental): Participants will be provided with A4i-O for one month.
  Interventions: Device: App for Independence-O (A4i-O)

INTERVENTIONS:
Device: App for Independence-O (A4i-O) — A4i-O is a digital health platform designed to support individuals with opioid use disorders. A4i-O will focus on providing education on treatment options, recovery navigation, social activation and connections to a range of resources. It aims to assist with fostering self-management and recovery through identifying risks for relapse, navigating urges/cravings, coping with shame/guilt, avoiding relapse, moving forward after relapse, and lived experiences. Daily wellness and goal attainment check-ins to highlight mental health trajectories will be prompted. With appropriate consent from both the client and provider, a provider dashboard is accessible to the client's provider prior to their appointment, generating a summary of day-to-day wellness ratings, responses to reminders, goal progressions, and other self-reported measures from the platform.

SUMMARY:
For the purposes of beta testing the first version of A4i-O, 15 individuals with OUD will use the platform for one month. From a design perspective this sample size is viewed as being sufficient to answer questions regarding app functionality and feasibility before moving to larger trials. Additionally, 15 individuals is a larger sample size than in the A4i pilot. This is an open label pilot with a primary objective of troubleshooting and providing early feedback on the beta version of the technology. To that end, 15 participants are anticipated to be sufficient to provide robust, early feedback. As with the focus groups, through sampling an effort will be made to secure a diverse group. Any individuals who might be declined in that effort at this stage (e.g., it is determined that no more male identifying participants are needed but they were interested) would be invited to take part in the subsequent RCT.

DETAILED DESCRIPTION:
Recruitment

Recruitment will be conducted through several mechanisms. First, with permission to do so by their clients, clinicians from within and external to CAMH are able to refer their clients to the study by emailing the study team. Participants recruited from Component 1 will be presented with the opportunity to participate in Component 2 via phone call. Clinicians will be made aware of the study via phone call. Potential service provider participants will be approached after they have been identified by the OUD participants who have formally consented to providers being asked to participate with them. Recruitment posters will be sent out to existing partnerships outlined in the component 1 portion of the protocol using the email templates provided. Second, component 2 will leverage the CLEARR recruitment strategy already approved and implemented in the COMPASS outpatient program at CAMH. CLEARR will be used to recruit participants for this research study. All new referrals will be reviewed by the CLEARR coordinator and CLEARR physician for eligibility to participate using minimal inclusion/exclusion criteria outlined. Once a patient is identified as potentially suitable for the research study, the attending physician will be notified via outlook calendar invite or email that their patient may be eligible for the research study. The attending physician will decide whether research is appropriate for the patient and if so, they will ask the patient for consent to be contacted regarding the research study. If the patient provides verbal consent to be contacted to receive more information about the research study, the physician will connect the patient with the CLEARR coordinator or research team who will further explain the research study. No personal health information (PHI) will be given to the research team prior to obtaining the patient's consent. The investigators have attached the letter of approval and the approved protocol to this submission. As part of the CLEARR protocol, willing participants will be pre-screened by a program RA and provided with study options/opportunities to participate based on self-reported criteria. No access to EMR prior to study consent is required for this process. Below is language provided by the SUHR centralized program:

The Substance Use Health Research (SUHR) Centralized Recruitment Database will be used to recruit participants for this study. Designated Research Personnel (DRP) or Study Specific Research personnel will prescreen individuals to support triaging and referral of individuals to prospective studies. Once a potential participant has been triaged, DRP will send preferred contact information to the Study Specific Research personnel who will reach out to the individual to further explain the study. Responses will be passed to the Study Specific Research Personnel only with the potential participant's consent.

Consent Process

Participants will be provided with a clear explanation of the objectives, procedures, risks and benefits of the study and all questions will be answered. Questions will be asked of subjects to ensure that they understand the nature of the research, the risks and potential benefits of study participation, and their rights as research subjects prior to obtaining their signature on the informed consent document. Participants will be informed of their responsibility to tell the research team of any medical conditions, medications, and changes in their health (e.g. pregnancy) while participating in this study. The PI will be consulted if the research analyst has any concerns about the participant's ability to understand any study procedures. Participant understanding will be assessed by the RA using a post-consent discussion quiz about key procedures in the study. If participant can recall and explain most of the procedures they will be asked if they would like to provide consent. If participants understand only the minority of procedures, the PI will be consulted. The PI will discuss the situation with the RA and, based on that conversation, may connect with the prospective participant to follow up and assess further. If it is decided that the individual is not capable of consenting, they will be thanked for their interest and informed that the investigators can't proceed with their participation as they appear to be struggling to understand what is involved. The investigators will not be formally assessing language comprehension or learning disability. The assessment will be based upon their demonstrated ability to understand the conditions of consent and the nature of the study. With participant permission, their clinicians may also be consulted to better understand the participant's capacity to provide consent. The RA may share with the participant's clinician the amount and type of information the participant seemed to have difficulty remembering or understanding from the consent form. In response, the study team will seek to investigate whether the participant's clinician has any concerns with the participant's capacity to understand or provide consent. As consent is an ongoing process, the investigators will continue to educate participants about the nature of the research and address any questions that may arise throughout the course of the study.

Assessments

Assessments will be scheduled via email and/or telephone by the study RP. All assessments will be conducted either virtually (via WebEx using either the teleconferencing or videoconferencing features depending on the participant's preference) or in person (onsite at the CAMH Queen Site). If they choose the virtual option, participants will be provided with the meeting link and phone number to join the WebEx call. The study RP will also use screen sharing to show the participant the questionnaires to assist with completing the assessment. If they choose in person, the person will be provided instructions to the CAMH Queen Site where the RP will meet them by the screening station to bring to the room that the research personnel has booked. The RP will then provide a CAMH approved tablet.. Participants will have the option to complete some brief (non-clinical) surveys over email, in the event of technical difficulties or time constraints. These surveys include the participant satisfaction survey. Survey responses will be secured using REDCap software. REDCap is a software located on Secure CAMH networks, the survey is not accessible or editable by external link once the survey is completed. So, if anyone intercepted the email with a link after the participant filled out the survey the information captured in the survey would not be accessible.

Interviews

Semi-structured interviews will be recorded using WebEx and transcribed verbatim. Transcripts are automatically provided by WebEx when the recording function is used. Within 30 days the recording will be deleted from WebEx and will be stored on the T-Drive. The study staff conducting the focus groups will review the recording and correct any mistakes in the transcript that may have occurred during automated transcription. Following transcription, the video will be deleted, and no identifiable information will be included in the transcripts.

A4i-O Installation

Installations will be conducted after the screening/baseline assessment either virtually (via WebEx using either the teleconferencing or videoconferencing features depending on the participant's preference) or in person (across from each other on-site following proper COVID safety protocols). Although there is no app user manual, participants will receive thorough instructions on how to use the app when on-boarded and can use the navigational tools within the app shown in Appendix 7. As well, a staff member will check-in with the participant within their first week of using the app to troubleshoot for any technical difficulties the participant may be experiencing. The RP conducting the installation will walk the participant through the installation and how to use the app by showing the participant (either a screen share or on their own device) what they app looks like and how to use each feature.

First Week Check-Ins

At the end of the first week, participants will be contacted for a brief check in about their experience with the app to see if they are having any challenges using the technology. Problems will be addressed by study staff as soon as possible.

Provider Dashboard Summaries

Anonymized summaries of the dashboard data will be sent to providers monthly via password protected files. Providers will also be able to log in to view the dashboard through the A4i-O portal. In the current version of A4i the dashboard summaries include user-entered information on mood ratings, reported sleep quality, medication adherence, and goal progression. The exact information available through the dashboard in Component 2 may be subject to change based on the results of Component 1. The intended use of the portal is to help clinicians have a better understanding of these variables in their client's lives outside appointments. Clinicians are instructed to use this information to inform their care if and how they see clinically fit. Clinicians can access these summaries through the clinical portals at any time. Participants are advised that the app is not to be used as a means of contacting their clinicians with the expectation of a response.

Data Analysis

Interview recordings will be transcribed verbatim. The content of the interviews will be thematically analysed with a consensus process used to validate the analysis (1). Quantitative analyses will be primarily descriptive, with outcomes probed (with sample size caveats) using paired samples t-tests and Cohen's d effect size analyses.

Conflict of Interest

In the interest of ensuring full disclosure, the A4i-O app is being developed together with a private company, A4i Inc. Both CAMH and Sean Kidd, the lead researcher, own and have shares in A4i. Sean Kidd holds a position as an officer of A4i as the co-founder and co-owner. Steps being taken to address this conflict of interest include things like disclosing this information whenever people are approached about research with A4i, having the data analyzed by experts not involved in A4i, and making anonymized data available for other researchers to examine and confirm.

ELIGIBILITY:
Inclusion Criteria:

1. Participants will be adults, 18 years of age or older, with a provider-assigned diagnosis of OUD confirmed by the SCID-5. Electronic medical records will be accessed for CAMH clients after informed consent is obtained to confirm the OUD diagnosis. For clients who were recruited externally and do not have a CAMH chart, confirmation of diagnosis will be sought from the referring clinician.
2. All participants will be engaged in outpatient psychiatric treatment for OUD.
3. All participants will currently be engaged in opioid agonist treatment.
4. Proficiency in English via ability to understand written/verbal communication during consent process. Any RA concerns about ability to understand English will be brought to the PI for determination of next steps (see consent procedures below).
5. Own and use an Android or iOS smartphone.
6. All participants will be open to having their care provider participate in the study

Exclusion Criteria:

1. Lack of capacity to consent.
2. Intellectual disability.
3. Experiencing distress at a level that would affect research and technology engagement (e.g., acute suicidality).

Criteria (service providers): Service providers will be psychiatrists and case managers engaged in the care of the participants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
A4i-O Total Time Used | 1 month
  Total time spent on the A4i-O app will be measured for each participant.
A4i-O Login Frequency | 1 month
  Number of times participants login to the A4i-O app will be calculated.
A4i-O Nature of Use Metrics | 1 month
  The frequency and type of A4i-O features used by each participant will be measured.
A4i-O Feedback from Participants and Providers | 1 month
  The Research Personnel will contact both providers and participants to complete a brief semi-structured interview assessing strengths (generally and in clinical interactions) and limitations of A4i-O and any risks not otherwise reported or observed during study operations.
Participant Satisfaction with A4i-O | 1 month
  Participant satisfaction with the technology will also be examined using the 26-item Acceptability/Usability Digital Health Technology scale used by Ben-Zeev and colleagues (2). Minimum values: -1, maximum values: 1, with a higher score indicating increased satisfaction (better outcome).
Safety and Critical Incidents | 1 month
  Safety will be assessed through information gathered via all study-related interactions with significant safety concerns operationalized as one or more critical incidents occurring in which there is evidence of an association between the incident and A4i-O use.

SECONDARY OUTCOMES:
General Symptom Severity | 1 month
  General symptomatology will be assessed using the 53-item, 5-point likert scale Brief Symptom Inventory. Minimum value: 0, and maximum value: 4, with higher scores indicating a worse outcome.
Substance Use Dependence | 1 month
  Specific to addictions, including opioids, the Severity of Dependence Scale will be used - for this trial altering the time period of reference from 2 months to 1 month (3). The SDS assesses subjective dependence to a range of substances with 5 item subscales answered using a 4-point likert response range. Minimum value: 0, and maximum value: 3, with higher scores indicating a worse outcome.
Treatment Engagement | 1 month
  Treatment Engagement will be measured using (i) the 4-item Brief Adherence Rating Scale (4) with responses obtained by both providers and participants to assess medication adherence. Minimum value: 1, and maximum value: 4, with higher scores indicating higher medication adherence (better outcome).
General Adherence to Treatment | 1 month
  The 5-item, 6-point likert scale Medical Outcomes Study general adherence scale (5) to capture broader adherence to treatment recommendations (again triangulated with provider responses) will be assessed. Minimum value: 1, and maximum value: 6, with higher scores indicating higher general adherence (better outcome).

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
If the results of this study are published, participant's identity will remain confidential. It is expected that the information collected during this study will be used in analyses and published to the scientific community at meetings and in journals. With participant consent, de-identified data from this study may be shared with the research community at large to advance science and health. The investigators will remove or code any personal information that could identify participants before files are shared with other researchers to ensure that by current scientific standards and known methods, no one will be able to identify participants from the information the investigators share.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Hsieh HF, Shannon SE. Three approaches to qualitative content analysis. Qual Health Res. 2005 Nov;15(9):1277-88. doi: 10.1177/1049732305276687. PMID 16204405
- [Background] Ben-Zeev D, Brenner CJ, Begale M, Duffecy J, Mohr DC, Mueser KT. Feasibility, acceptability, and preliminary efficacy of a smartphone intervention for schizophrenia. Schizophr Bull. 2014 Nov;40(6):1244-53. doi: 10.1093/schbul/sbu033. Epub 2014 Mar 8. PMID 24609454
- [Background] Derogatis, L.R.(1993). BSI Brief Symptom Inventory: Administration, Scoring, and Procedure Manual (4th Ed.). Minneapolis, MN: National Computer Systems.
- [Background] Byerly MJ, Nakonezny PA, Rush AJ. The Brief Adherence Rating Scale (BARS) validated against electronic monitoring in assessing the antipsychotic medication adherence of outpatients with schizophrenia and schizoaffective disorder. Schizophr Res. 2008 Mar;100(1-3):60-9. doi: 10.1016/j.schres.2007.12.470. Epub 2008 Feb 5. PMID 18255269
- [Background] Sherbourne CD, Hays RD, Ordway L, DiMatteo MR, Kravitz RL. Antecedents of adherence to medical recommendations: results from the Medical Outcomes Study. J Behav Med. 1992 Oct;15(5):447-68. doi: 10.1007/BF00844941. PMID 1447757